CLINICAL TRIAL: NCT00487318
Title: A Randomized Controlled Trial of Adding Fluvastatin to Standard Medical Treatment (SMT) and a Pilot Trial of Rosuvastatin and Other Statins With SMT, for Patients Infected With Chronic Hepatitis C Who Are Naive to Therapy.
Brief Title: Fluvastatin, Rosuvastatin Added to Pegylated Interferon and Ribavirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bader, Ted, M.D. (Individual)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ted Bader, MD, Director of Liver Diseases, VA Medical Center, Bader, Ted, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13358
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Hepatitis C
Keywords: fluvastatin; hepatitis C; chronic hepatitis C; not previously treated with pegylated interferon and ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Standard of Care; Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Plus statin (Experimental): The addition of fluvastatin or rosuvastatin or other statins to the standard of care of peginterferon and ribavirin.
  Interventions: Drug: fluvastatin
- 2 (Active Comparator): Administration of the standard of care for hepatitis C of peginterferon and ribavirin.
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: standard of care — peginterferon/RBV
  Arms: 2
Drug: fluvastatin — Add fluvastatin at 20-40 mg/day to standard of care
  Other Names: Lescol
  Arms: Arm 1 Plus statin

SUMMARY:
Hypothesis: addition of fluvastatin will increase the cure rate of standard anti-HCV therapy. Summary: This trial is limited to veterans in Oklahoma who qualify for care with the Veterans Administration. It is a randomized control format including genotypes 1 and 3. There will also be pilot arms for HCV carriers who present for screening already on a statin, who will be allowed to stay on their current statin or switched to another statin. In all ways, standard therapy as noted on pegylated interferon and ribavirin will be given per FDA package insert.

ELIGIBILITY:
Inclusion Criteria:

* Not previously treated.
* Off alcohol and marijuana for 6 months
* HCV RNA positive

Exclusion Criteria:

* HIV positive
* Advanced liver disease
* Advanced cardiopulmonary disease
* Chronic renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Sustained Viral response | 72 weeks

SECONDARY OUTCOMES:
Viral load at 4, 12 and 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ted F Bader, MD, Principal Investigator — OUHSC and VAMC
Locations (1):
- Veterans Administration Medical Center, Oklahoma City, Oklahoma, United States